CLINICAL TRIAL: NCT03761615
Title: Observational Study of Patient Important Outcomes in Pregnant Patients With Type 1 Diabetes Mellitus on Insulin Pump
Brief Title: Longitudinal Observation of Insulin Requirements and Sensor Use in Pregnancy
Acronym: LOIS-P
Status: Completed | Type: Observational
Sponsor: Sansum Diabetes Research Institute (Other)
Collaborators: Harvard University (Other); Mayo Clinic (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 18-007081
Record Dates: First submitted 2018-11-24; First posted 2018-12-03 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes Mellitus; Pregnancy in Diabetics
Keywords: type 1 diabetes; pregnancy; continues glucose monitoring; artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Pregnancy in Diabetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- type 1 diabetes and pregnancy: Pregnant women with T1D on insulin pumps (CSII/SAP/PLGS) will be offered enrollment in a prospective study that will capture: 1) Dexcom G6 CGM data, 2) self-monitoring of blood glucose (SMBG), 3) insulin pump settings, 4) insulin delivery records, and 5) maternal and fetal outcomes.
  Interventions: Device: Dexcom G6 CGM

INTERVENTIONS:
Device: Dexcom G6 CGM — All women in the study will be given Dexcom G6 CGM and a study glucometer.

SUMMARY:
The overall goal of this study is to enroll pregnant women with type 1 diabetes and follow their glycemic outcomes prospectively throughout pregnancy and into the post-partum period. The investigators anticipate that when compared to subjects using an Artificial pancreas system (AP) as part of a future protocol, this comparator group of subjects undergoing usual care will exhibit less time in target continuous glucose monitoring (CGM) glucose range defined as 63-140 mg/dL and an increased duration of hypoglycemia with CGM glucose <63 mg/dL.

DETAILED DESCRIPTION:
This is an observational study. Data collected will include records of continuous glucose monitoring (CGM) based glucose, insulin delivery, self-monitoring of blood glucose (SMBG), and maternal and fetal outcomes from pregnant women with type 1 diabetes. These data will be used to: (1) develop and refine algorithms for an AP system tailored to the needs of pregnant women with type 1 diabetes, (2) to serve as a comparator group for concurrent AP protocols, (3) describe Dexcom G6 CGM data throughout the pregnancy, and (4) describe insulin changes which occur in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis, based on investigator assessment, of T1D for at least one year and using insulin for at least 1 year.
* Criteria for documented hyperglycemia (at least 1 must be met):

  * Fasting glucose ≥126 mg/dL
  * Two-hour OGTT glucose ≥200 mg/dL
  * HbA1c ≥6.5% documented
  * Random glucose ≥200 mg/dL with symptoms
  * No data at diagnosis is available but the participant has a convincing history of hyperglycemia consistent with T1D
* Criteria for requiring insulin at diagnosis (1 must be met):

  * Participant required insulin at diagnosis and continually thereafter.
  * Participant did not start insulin at diagnosis but upon investigator review likely needed insulin (significant hyperglycemia that did not respond to oral agents) and did require insulin eventually and used continually.
  * Participant did not start insulin at diagnosis but continued to be hyperglycemic, had positive islet cell antibodies - consistent with latent autoimmune diabetes in adults (LADA) and did require insulin eventually and used continually.
* Currently using an insulin pump for diabetes management
* Currently using or willing to use an insulin-to-carbohydrate ratio to calculate meal bolus sizes
* Willing to change insulin infusion site at least every 3 days.
* Confirmed pregnancy
* Current gestational age <17 weeks
* Age 18-40 years
* HbA1c <10.0%
* Demonstration of proper mental status and cognition for the study
* Ability to access the internet and upload CGM data remotely if needed
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* 670 G users in Auto mode
* Current gestational age ≥17 weeks
* Cystic fibrosis
* A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

  * Inpatient psychiatric treatment in the past 6 months
  * Abnormal renal function test results (calculated GFR <60 mL/min/1.73m2); testing required for subjects with diabetes duration of greater than 5 years post onset of puberty
  * Active gastroparesis
  * Abuse of alcohol or recreational drugs
  * Infectious process not anticipated to resolve prior to study procedures (e.g. meningitis, pneumonia, osteomyelitis)
  * Uncontrolled arterial hypertension (Resting diastolic blood pressure >95mmHg and/or systolic blood pressure >160 mmHg) at the time of screening
  * Chronic oral steroid use
* A recent injury to body or limb, muscular disorder, use of any medication, any carcinogenic disease, or other significant medical disorder if that injury, medication or disease in the judgment of the investigator will affect the completion of the protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women 18 years of age or older with T1D using an insulin pump
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Dassau, PhD, Principal Investigator — Harvard University; Carol Levy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Yogish C Kudva, MD, Principal Investigator — Mayo Clinic; Jordan E Pinsker, MD, Principal Investigator — Sansum Diabetes Research Institute; Barak Rosenn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kristin Castorino, DO, Principal Investigator — Sansum Diabetes Research Institute; Grenye O'Malley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Plan to create a public database of study results per NIH open data policy.
Supporting Information: Study Protocol, SAP
Time Frame: 1 year after study data analysis is complete and results are published.

REFERENCES:
- [Result] O'Malley G, Ozaslan B, Levy CJ, Castorino K, Desjardins D, Levister C, McCrady-Spitzer S, Church MM, Kaur RJ, Reid C, Kremers WK, Doyle FJ, Trinidad MC, Rosenn B, Pinsker JE, Kudva YC, Dassau E. Longitudinal Observation of Insulin Use and Glucose Sensor Metrics in Pregnant Women with Type 1 Diabetes Using Continuous Glucose Monitors and Insulin Pumps: The LOIS-P Study. Diabetes Technol Ther. 2021 Dec;23(12):807-817. doi: 10.1089/dia.2021.0112. Epub 2021 Aug 17. PMID 34270347
- [Result] Kaur RJ, Smith BH, Ozaslan B, Pinsker JE, Trinidad MC, O'Malley G, Desjardins D, Castorino KN, Levister C, Reid C, McCrady-Spitzer S, Ogyaadu SJ, Church MM, Piper M, Kremers WK, Rosenn B, Doyle FJ 3rd, Dassau E, Levy CJ, Kudva YC. Hypoglycemia in Prospective Multicenter Study of Pregnancies with Pre-Existing Type 1 Diabetes on Sensor-Augmented Pump Therapy: The LOIS-P Study. Diabetes Technol Ther. 2022 Aug;24(8):544-555. doi: 10.1089/dia.2021.0479. PMID 35349353

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Type 1 Diabetes and Pregnancy
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Pregnant women with preexisting T1D for at least 1 year were enrolled before 17 weeks gestational age.
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.2 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Gestational Age at Enrollment [Mean (Standard Deviation); unit: weeks] | 11.2 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Range Glucose Levels 63-140 mg/dL as Determined by CGM
Description: Time in range defined as 63-140 mg/dL as determined by CGM analysis
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
percentage of time | 59 (14)

2. Secondary Outcome: Percentage of Percentage of Time Spent Below Target Glucose (<63 mg/dL) as Determined by CGM
Description: Time spent below target cgm glucose range defined as glucose <63 mg/dL
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
percentage of time | 3 (3)

3. Secondary Outcome: Percentage of Time Spent Above Target Glucose Range (> 140 mg/dL) as Determined by CGM
Description: Time spent above target cgm glucose range defined as >140 mg/dL
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
percentage of time | 38 (15)

4. Secondary Outcome: Episodes of Clinically Significant Hyperglycemia
Description: Episodes of clinically significant hyperglycemia with CGM glucose >180 mg/dL
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
episodes | 0.08 (0.28)

5. Secondary Outcome: Total Daily Insulin Requirements Over Last 2 Weeks of Third Trimester
Description: Total daily insulin requirements (units/kg/day) over last 2 weeks of third trimester
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
units/kg/day | 0.88 (0.04)

6. Secondary Outcome: Basal Insulin Requirements Over Last 2 Weeks of Third Trimester
Description: Basal daily insulin requirements (units/kg/day) over last 2 weeks of third trimester
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units/kg/day
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
units/kg/day | 0.4 (0.03)

7. Secondary Outcome: Carbohydrate Consumption Over Last 2 Weeks of Third Trimester
Description: Carbohydrate consumption (g/(kg*day)) over last 2 weeks of third trimester
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: g/(kg*day)
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
g/(kg*day) | 1.76 (0.11)

8. Other Pre Specified Outcome: Ketoacidosis
Description: Episodes of ketoacidosis requiring emergency room or hospital admission
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: events during pregnancy
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
events during pregnancy | 0.0 (0.0)

9. Other Pre Specified Outcome: Maternal Complications
Description: Maternal complications including preeclampsia, pregnancy induced hypertension and polyhydramnios
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: complications
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
complications | 0.36 (0.49)

10. Other Pre Specified Outcome: Gestational Weight Gain
Description: Gestational weight gain each week
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Measure: Mean (Standard Deviation); unit: kg/week
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
kg/week | 0.42 (0.14)

11. Other Pre Specified Outcome: Gestational Age at Delivery
Description: Gestational age at delivery (Weeks)
Time Frame: Immediately at birth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
weeks | 37.7 (1.6)

12. Other Pre Specified Outcome: Birth Weight of Baby
Description: Birth weight of baby (kg)
Time Frame: Immediately at birth
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
grams | 3700 [2135 to 4345]

13. Other Pre Specified Outcome: LGA
Description: Number of Large for Gestational Age based on WHO criteria at time of delivery
Time Frame: Immediately at birth
Population: Infants delivered
Measure: Count of Participants; unit: Participants
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
Participants | 14

14. Other Pre Specified Outcome: Preterm Birth
Description: Number of infants born late preterm birth (at 34-37 weeks)
Time Frame: Immediately at birth
Population: Number of infants delivered preterm late preterm (at 34-37 weeks).
Measure: Number; unit: infants
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
infants | 8

15. Other Pre Specified Outcome: Neonatal NICU Stay
Description: Number of infants requiring neonatal NICU stay
Time Frame: Prior to 17 weeks gestation (enrollment) through up to 6 weeks postpartum
Population: Number of infants admitted to NICU
Measure: Number; unit: infants
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
infants | 10

16. Other Pre Specified Outcome: Cesarean Delivery
Description: Number of participants that underwent primary cesarean section for delivery
Time Frame: Immediately at birth
Measure: Count of Participants; unit: Participants
Arm/Group | Type 1 Diabetes and Pregnancy
Number analyzed (Participants) | 25
Participants | 13

ADVERSE EVENTS:
Time Frame: During pregnancy, up to 39 weeks
Arm/Group | Type 1 Diabetes and Pregnancy
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 9/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 1 Diabetes and Pregnancy (N=25)
Severe Hypoglycemia (Endocrine disorders) | 2 (2) — Severe hypoglycemia with possible seizures
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 1 Diabetes and Pregnancy (N=25)
gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 5 (5)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT03761615/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/15/NCT03761615/ICF_001.pdf